CLINICAL TRIAL: NCT06089343
Title: Exploring the High-risk Features of Coronary Lesions Using CT Angiography and Optical Coherence Tomography
Brief Title: High-risk Features of Coronary Lesions in CTA and OCT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ACS-CTA&OCT
Record Dates: First submitted 2023-10-13; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culprit: Plaques which is related with acute coronary syndrome
  Interventions: Diagnostic Test: Coronary CT angiography
- Non-culprit: Plaques which is not related with acute coronary syndrome
  Interventions: Diagnostic Test: Coronary CT angiography

INTERVENTIONS:
Diagnostic Test: Coronary CT angiography — Comprehensive hemodynamic and plaque features derived from CTA and verified by OCT of all culprit and non-culprit lesions to predict ACS.

SUMMARY:
This study is a multicenter and retrospective study. ACS patients who underwent CCTA or OCT from 1 months to 3 years prior to the event will be retrospectively identified. Plaques in the non-culprit vessels will be regarded as a primary control group.

DETAILED DESCRIPTION:
The high-risk features of plaque rupture and subsequent acute coronary syndrome (ACS) are not fully identified. Plaque features, hemodynamic forces, and the interaction between these factors may cause plaque instability and subsequent clinical events. A previous study showed that the addition of hemodynamic parameters calculated noninvasively from coronary computed tomography (CCTA) using computational fluid dynamics (such as wall shear stress and axial plaque stress) improved the ability to predict the risk of ACS compared with conventional approaches based on anatomical stenosis severity and adverse plaque characteristics. Wall shear stress and axial plaque stress derived from CT were highly correlated to those derived from optical coherence tomography (OCT). In addition, other hemodynamic parameters, such as oscillatory shear index, endothelial shear stress (ESS), and spatial ESS gradient have also been demonstrated to be associated with unstable plaque. In this regard, we designed this study to find the best hemodynamic and plaque features derived from CTA and verified by OCT to predict ACS, and to investigate whether a comprehensive risk prediction model with them has an incremental value in a larger population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who presented with ACS and underwent invasive coronary angiography or OCT
2. The patients who underwent coronary CT angiography, regardless of the reason (for example, routine healthcare check-up, or evaluation for stable angina or atypical chest pain) prior to the acute event.
3. Time limit of CCTA: 1 months ~ 3 years prior to the event.

   * Exclusion Criteria:

Patients with stents in two or more vessel territories prior to CCTA Poor quality of CCTA which is unsuitable for plaque and CFD analysis Patients with ACS culprit lesion in a stented segment Patients with previous history of coronary artery bypass graft surgery Patients with revascularization after CCTA and before ACS event Secondary ACS due to other general medical conditions, such as sepsis, arrhythmia, bleeding, etc.

--Additional exclusion criteria for Computational Fluid Dynamics Poor quality CCTA images unsuitable for CFD and plaque analysis No unprocessed CCTA data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented with acute coronary syndrome (acute myocardial infarction or unstable angina) and had undergone CCTA from 1 months to 3 years prior to the event.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
discrimination index of prediction model | 1 months - 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China